CLINICAL TRIAL: NCT05241132
Title: Tislelizumab Combined With Chemotherapy in the Treatment of Bone Metastases of Unknown Primary: A Prospective, Open-label, Single-arm Clinical Study
Brief Title: Tislelizumab Combined With Chemotherapy in the Treatment of Bone Metastases of Unknown Primary
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Wei Xu, Professor of Orthopaedic department of Changzheng Hospital, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021SL047
Record Dates: First submitted 2022-01-23; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Cancer of Unknown Primary; Bone Cancer Metastatic; Tislelizumab; Gene Mutation-Related Cancer; Immune Evasion, Tumor; Chemotherapy Effect
Keywords: Bone metastases from cancer of unknown primary; Cancer of unknown primary; Tislelizumab; Chemotherapy Effect; Immunotherapy; Gene expression spectrum
MeSH Terms: conditions — Neoplasms | interventions — tislelizumab; Drug Therapy; Cisplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, open phase II clinical study
Masking Description: Prior to enrollment in the study, doctors asked and recorded the patient's medical history, and if eligible participants volunteered to participate in the study, they would sign informed consent.If they are not willing to participate in the study, we will do the usual treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BMCUP treated with Tislelizumab and chemotherapy (Experimental): Patients with bone metastases from cancer of unknown primary (BMCUP) diagnosed according to the criteria defined in the 2015 European Society of Medical Oncology (ESMO) clinical Practice Guidelines and with bone metastases confirmed by imaging and histology that cannot be completely resected
  1. Cisplatin: 100mg/m2, injected intravenously every 3 weeks, 8 cycles (period 21 days)
  2. Paclitaxel (albumin-bound) : paclitaxel, 175mg/m2, given intravenously every 3 weeks for 8 cycles (period 21 days).
  3. Tislelizumab: 200mg, given intravenously every 3 weeks until disease progression or unacceptable toxicity or death or subject withdrawal of informed consent.
  Interventions: Drug: Tislelizumab plus chemotherapy

INTERVENTIONS:
Drug: Tislelizumab plus chemotherapy — 1. Cisplatin: 100mg/m2, injected intravenously every 3 weeks, 8 cycles (period 21 days)
  2. Paclitaxel (albumin-bound) : paclitaxel, 175mg/m2, given intravenously every 3 weeks for 8 cycles (period 21 days).
  3. Tislelizumab: 200mg, given intravenously every 3 weeks until disease progression or unacceptable toxicity or death or subject withdrawal of informed consent.
  Other Names: Cisplatin; Paclitaxel

SUMMARY:
Through scientific and rigorous design, implementation, follow-up and statistics, the sponsor aims to explore the clinical efficacy and safety of Tislelizumab combined with chemotherapy (platinum + paclitaxel) in the treatment of patients with bone metastases cancer with unknown primary, and provide a better treatment plan for these patients.

1. Primary outcome: Objective response rate (ORR)
2. Secondary outcomes: disease control rate (DCR), duration of remission (DOR), progression-free disease (PFS), overall survival (OS), median PFS, median OS, stratification based on clinical features and PD-L1 expression, adverse reactions (AEs), and quality of life.

DETAILED DESCRIPTION:
Unknown primary metastatic carcinoma is a general term for independent metastatic tumors, which are histologically confirmed as metastatic carcinoma but whose primary anatomic site cannot be determined after examination. It accounts for about 3% ~ 5% of all new cancers in humans, and is the 7th ~ 8th most common malignant tumor and the 4th most common fatal cancer in humans.CUP is typically characterized by aggressive and early metastasis and unpredictable metastasis. The disease is not a single disease, but a heterogeneous collection of tumors composed of different primary tumor types that cannot be recognized Bone is the third most common site of CUP, and bone metastases from cancer of unknown primary (BMCUP) is a type of CUP with poor overall prognosis. The primary site of the tumor was determined. BMCUP is a type of heterogeneous tumor with bone metastases confirmed by biopsy but whose primary anatomic site cannot be determined after detailed history, physical examination and relevant experimental examination.BMCUP accounts for about 10% of CUP, which is common in adults with a median onset age of 65-90 years and slightly more in men than women.The spine is the most common site of BMCUP, followed by the pelvis and long bones.Adenocarcinoma was the main pathologic type of BMCUP, with low and medium differentiated adenocarcinoma (64%), undifferentiated carcinoma (20%), neuroendocrine carcinoma (9%) and squamous cell carcinoma (7%).Patients with BMCUP usually have a poor prognosis, with an average survival of 3 to 12 months.

Currently, empire-based chemotherapy, including platinum and taxanes, is still the main treatment for CUP and BMCUP, but the effect is not ideal and the survival rate is very low (median overall survival, about 6-9 months).In recent years, gene expression profiling is a new diagnostic technique, which makes it possible to predict the origin of tumor tissue based on the expression profiling of specific sites. Several of these molecular profiling methods, including reverse transcription polymerase chain reaction (RT-PCR) analysis and DNA microarray analysis, have been developed to trace the primary foci of CUP and BMCUP. In addition, the results of gene expression profiling can indicate the information of tumor genetic abnormalities and thus potential targeted drugs. However, Hayashietal etal., published in JCO in 2019, concluded that "although the prediction of the primary site seems to have prognostic value,However, cuP-site-specific therapy based on microarray mapping did not result in a significant improvement in 1-year survival compared with empirical platinum-paclitaxel therapy ". At present, the systemic treatment of CUP and BMCUP is still not ideal, and finding new effective and safe drug treatment is the key research content of this kind of disease.

In recent years, with the deepening of the research on the regulation mechanism of the immune system and the emergence of immune checkpoint inhibitors, biological therapy with tumor immunotherapy as the core has developed rapidly, and now has become another major cancer treatment mode after chemotherapy and targeted drugs. When the body encounters cancer cells, antigen presenting cells (APC) capture antigen (Ag) and present it to T cells. After activation of T cells, programmed cell death protein 1 (PD-1) receptor can be expressed in T cells and transmit negative regulatory signals to T cells by binding to PD-L1 ligand on tumor cells and APC surface, thus inhibiting the immune response. Immune checkpoint inhibitors block the binding of the PD-1 receptor to the PD-L1 ligand, thereby enhancing the anti-tumor immune response.Pd-1 and PD-L1 inhibitors play a significant antitumor effect in lung cancer, melanoma, kidney cancer and other malignant tumors, but there are no literature reports on the efficacy and safety of immune checkpoint inhibitors in CUP and BMCUP. According to the search results of our treatment group, ClinicaTtrails. Gov has registered clinical trials under research, and the studies related to the application of immune checkpoint inhibitors in CUP include Tom Baker Cancer Center in Canada, a prospective single-arm study of paprizumab monotherapy in CUP patients with poor prognosis, which is still recruiting patients.

Tislelizumab is a humanized IgG4 monoclonal antibody against PD-1, which is an "immune checkpoint" inhibitor. It can bind to the PD-1 receptor on the cell surface and block the binding of PD-L1 and PD-L2. Thus, the escape state of tumor immunity is reversed and the killing activity of T cells is restored. Compared with other PD-1 antibodies, Tislelizumab can reduce the binding of FcγR on macrophages, thereby reducing antibody-dependent phagocytosis and possibly improving the resistance of PD-1 antibodies. It was approved for market in China on December 26, 2019. For the treatment of patients with recurrent or refractory classic Hodgkin's lymphoma, urothelial carcinoma, non-small cell lung cancer, hepatocellular carcinoma. In terms of safety, the most common grade 3 or higher adverse reactions associated with Tislelizumab were elevated glutamyltransferase, anemia, and glutamic-oxalacetic transaminase.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent/consent for the trial.
2. Be at least 18 years old on the day of signing the informed consent.
3. Patients with bone metastases from cancer of unknown primary (BMCUP) diagnosed according to the criteria defined in the clinical practice guidelines of the European Society of Medical Oncology (ESMO) in 2015 and confirmed by imaging and histology to have bone metastases that cannot be completely resected.
4. Did not receive systemic treatment.
5. Have at least one measurable lesion according to RECIST1.1, willing to agree to archived tumor (in formalin fixed paraffin-embedded (FFPE) block) or fresh tumor material (cryogenic refrigerator or liquid nitrogen storage).
6. ECOG performance level 0 or 1 point.
7. The expected survival time is ≥3 months.
8. Adequate organ and bone marrow functions (all screening tests should be performed within 10 days of the start of treatment) :A) Absolute neutrophil count ≥1.5x109 /L.B) Platelet ≥100x109 /L.C) Hemoglobin ≥9g/dL(≥90g/L).D) No blood transfusion or erythropoietin dependence (within 7 days of evaluation).E) Serum creatinine ≤1.5x upper normal limit (ULN) or creatinine level > 1.5xULn, creatinine clearance ≥60 ml/min (creatinine clearance should be calculated according to institutional criteria).F) Patients with serum total bilirubin ≤1.5xULN or total bilirubin level > 1.5ULN, direct bilirubin ≤ULN.G) Aspartate aminotransferase ≤2.5xULN(if liver metastasis is present).H) Alanine aminotransferase ≤2.5xULN(if liver metastasis is present).I) Albumin ≥2.5g/dL.J) International standardized ratio (INR) or prothrombin time ≤1.5xULN(if subject is being treated with anticoagulant, prothrombin time or partial prothrombin time should be within the range expected for treatment with anticoagulant).K) Activated partial thrombin time ≤1.5xULN(prothrombin time or partial prothrombin time should be within the expected therapeutic range of anticoagulant use).L) Women with reproductive potential should undergo a mandatory serum-negative pregnancy within 72 hours prior to receiving the first dose of the study drug.M) Fertile female subjects must be willing to use appropriate contraceptive methods during the study up to 120 days after the last use of the study drug.Note: Abstinence is acceptable if this is the subject's usual lifestyle and preferred method of contraception.N) Male subjects with reproductive potential must consent to use appropriate contraceptive methods from the first study treatment until 120 days after the last study treatment.

Exclusion Criteria:

1. Unknown primary lesion of squamous cells.
2. in suspected lymphoma (e.g., leukocyte common antigen staining), malignant melanoma (for example, according to dye and beta hCG), gonads germ cell tumor (such as AFP and human chorionic gonadotropin), sarcoma (such as cell keratin and vimentin staining), neuroendocrine tumor (such as chromaffin granulocyte and synaptic staining).And male prostate cancer (e.g., prostate specific antigen staining).
3. apply to specific treatment, the patients of group (for example, only axillary lymph node metastasis of adenocarcinoma patients, peritoneal papillary serous carcinoma patients, only involving the neck, or groin lymph nodes of patients with squamous cell carcinoma, prompt germ cell tumors and beta hCG and/or AFP levels of patients with poorly differentiated carcinoma, and involves a single potentially resectable cancer patients).
4. Currently participating in and receiving study therapy, or participating in a study formulation and receiving study therapy or using study drug within 4 weeks of the first dose.
5. Confirmed immunodeficiency or receiving documented systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to receiving the first dose of tirelizumab.
6. Have active tuberculosis.
7. Have an allergic reaction to the study drug.
8. One has received radiotherapy within 14 days before the first treatment. If the subjects received radiotherapy, they must fully recover from the toxicity and / or complications caused by the intervention, according to the judgment of a qualified investigator, before starting the treatment.
9. Have received chemotherapy treatment.
10. Subjects must fully recover from surgery and related complications in the judgment of a qualified investigator prior to the initiation of treatment.
11. There is another known malignancy developing or requiring aggressive treatment.Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin, squamous cell carcinoma of the skin that has received potential treatment, or cervical carcinoma in situ.
12. Active central nervous system (CNS) metastases and/or cancerous meningitis are known.Brain metastasis treated subjects as long as they received in a stable condition (in the treatment of at least four weeks before the first trials there was no evidence of progress examined by CT or MRI brain, any neurological symptoms has returned to baseline), there was no evidence of brain metastases from new or expanded, and at least 7 days prior to treatment did not use steroids, can attend the test.This exception does not include cancerous meningitis, which is excluded regardless of clinical stability.
13. Active autoimmune disease requiring systematic treatment (i.e. disease improvers, corticosteroids, or immunosuppressants) within the past two years.
14. Having (noninfectious) pneumonia or a history of current pneumonia.
15. There is an active infection that requires systematic treatment.
16. History or current evidence of any condition, treatment or laboratory abnormality that is likely to confound the results of the study or interfere with the subject's participation throughout the study, or any history or evidence of any condition, treatment or laboratory abnormality that, in the opinion of a qualified investigator for the treatment, would not be in the subject's best interest to participate.
17. A known mental or substance abuse disorder interferes with compliance with test requirements.
18. The subject is pregnant or breast-feeding, or plans to become pregnant or a father during the expected duration of the trial, beginning with pre-screening or screening 120 calendar days after the last trial treatment and continuing 120 calendar days after the last trial treatment.
19. Once have received anti-PD-1, anti-PD-L1 or anti-PD-L2 preparation treatment.
20. A known history of human immunodeficiency virus (HIV).
21. Active hepatitis B (e.g., HBsAg reaction) or hepatitis C (e.g., detection of HCVRNA) is known.
22. Live vaccine should be administered within 30 calendar days of the planned initiation of study treatment.
23. Have a history of organ and/or bone marrow transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response(CR) and Partial Response(PR) in all participants according to RECIST,v1.1 | 3 years
  Proportion of patients whose tumor volume shrinks to a predetermined value and maintains the minimum time limit

SECONDARY OUTCOMES:
Disease control rate（DCR）according to RECIST,v1.1 | 3 years
  Proportion of patients whose tumors shrank or remained stable for a certain amount of time
Duration of remission (DOR) by Kaplan-Meier | 3 years
  The time between the first tumor evaluation for CR or PR and the first evaluation for PD (Progressive Disease) or death from any cause
Progression Free Survival (PFS) by Kaplan-Meier | 3 years
  The time span from the start of treatment to the onset of secondary growth
Overall survival (OS) by Kaplan-Meier | 3 years
  The time between randomization and the death of the patient from any cause
The median of Progression Free Survival (PFS) by Kaplan-Meier | 3 years
  Fifty percent of patients survival with respect to the The time span from the start of treatment to the onset of secondary growth
The median of overall survival (OS) by Kaplan-Meier | 3 years
  Fifty percent of patients survival with respect to The time between randomization and the death of the patient from any cause
Stratified analysis based on clinical features and PD-L1 expression | 3 years
  Stratified analysis
Adverse effects (AEs) according to NCI-CTCAE, v5.0 | 3 years
  The occurrence of adverse events was recorded
The quality of life according to QoF(sf-36) | 3 years
  Quality of life was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jianru Xiao, Profession, Study Chair — Chang Zheng Hospital; Wei Xu, Profession, Study Director — Chang Zheng Hospital; Bo Li, Profession, Principal Investigator — Chang Zheng Hospital; Hao Jiang, Doctor, Principal Investigator — Chang Zheng Hospital; Pengru Wang, Doctor, Principal Investigator — Chang Zheng Hospital
Locations (1):
- ChangZheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After completion
Supporting Information: Study Protocol
Time Frame: After completion
Access Criteria: 1111